CLINICAL TRIAL: NCT04973826
Title: A PHASE I, SINGLE CENTER, OPEN-LABEL STUDY TO ASSESS THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF AZTREONAM-AVIBACTAM ADMINISTERED AS SINGLE AND REPEATED INTRAVENOUS DOSES IN HEALTHY CHINESE PARTICIPANTS
Brief Title: Study to Assess the Pharmacokinetics, Safety and Tolerability of Aztreonam-Avibactam in Healthy Chinese Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C3601007
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: no clinically relevant abnormalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATM-AVI treatment arm (Experimental): Chinese healthy volunteers
  Interventions: Drug: Aztreonam-Avibactam

INTERVENTIONS:
Drug: Aztreonam-Avibactam — 500/167 mg ATM/AVI loading infusion, followed by 1500/500 mg ATM/AVI extended loading infusion, then 1500/500 mg ATM/AVI maintenance dose infusion every 6 hours

SUMMARY:
A Phase 1, single center, single arm, open-label study to assess the PK, safety and tolerability of Aztreonam-Avibactam after single and repeated IV infusion of doses in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male and female participants
* No clinical relevant abnormalities
* willing and able to comply with all study procedures
* BMI:17.5-30.5
* Sign informed consent

Exclusion Criteria:

* Any clinical significant illness
* History of alcohol abuse
* Use within 14 days prior the first study dose
* CL>80ml/min
* Abnormal vital signs, such 12-ECG, blood pressure and pulse rate
* Blood donation within 60days
* History of HIV, HBsAg, HBcAb, HCVAb
* Other medical or psychiatric may inappropriate for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3601007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 participants received assigned treatment of AZTREONAM-AVIBACTAM (ATM-AVI) and completed the treatment and follow-up phases.
Groups:
- AZTREONAM-AVIBACTAM (ATM-AVI): ATM-AVI was dosed in a fixed 3:1 ratio (ATM:AVI=3:1) in 12 healthy participants. On Day 1, participants received a 3-hour intravenous (IV) infusion of a single dose of 1500 mg ATM plus 500 mg AVI. On Day 2, participants received a loading (500 mg ATM plus 167 mg AVI infused over a 30-minute period)/extended loading dose (1500 mg ATM plus 500 mg AVI over a 3-hour period), followed by multiple maintenance doses of ATM-AVI IV infusion: 1500 mg ATM and 500 mg AVI were infused over 3 hours and administered every 6 hours (q6h) till morning of Study Day 4.
Period: Overall Study
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study medication.
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.08 (5.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 1 & 4 of Aztreonam
Description: Cmax was the maximum observed plasma concentration and was directly observed from data. Concentration values below the lower limit of quantification (LLQ) were set to zero. Geometric Mean analysis was on the log scale. Zero values were not included in geometric mean and geometric coefficient of variation calculation. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: The analysis population included all participants who received at least one dose of investigational product (ATM-AVI) and had at least one of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
micrograms per milliliter (ug/mL)
  Day 1 | 69.44 (15)
  Day 4 | 79.66 (12)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 1 & 4 of Avibactam
Description: as for outcome 1
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug/mL
  Day 1 | 13.93 (16)
  Day 4 | 14.03 (14)

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to 6 Hours (AUC6) on Day 1 of Aztreonam
Description: The area under the plasma drug concentration-time curve (AUC) was estimated from time 0 to 6 hours post dose. AUC6 was computed using the Linear/Log trapezoidal method. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/millilitre/hour (ng*hr/mL)
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
nanograms/millilitre/hour (ng*hr/mL) | 236.7 (14)

4. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to 6 Hours (AUC6) on Day 1 of Avibactam
Description: as for outcome 3
Time Frame: Post dose on day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ng*hr/mL | 42.36 (15)

5. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time of the Last Quantifiable Concentration (AUClast) on Day 1 & 4 of Aztreonam
Description: AUClast is area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL
  Day 1 | 287.8 (14)
  Day 4 | 336.4 (15)

6. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time of the Last Quantifiable Concentration (AUClast) on Day 1 & 4 of Avibactam
Description: as for outcome 5
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL
  Day 1 | 47.23 (15)
  Day 4 | 49.47 (18)

7. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to 24 Hours (AUC24) on Day 1 & 4 of Aztreonam
Description: AUC24 was defined as area under the plasma concentration-time profile from time zero to 24 hours post dose. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL
  Day 1 | 289.6 (14)
  Day 4 | 337.5 (15)

8. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to 24 Hours (AUC24) on Day 1 & 4 of Avibactam
Description: as for outcome 7
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL
  Day 1 | 47.33 (15)
  Day 4 | 49.47 (18)

9. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) on Day 1 & 4 of Aztreonam
Description: AUCinf was defined as area under the plasma concentration-time curve from time zero to infinity. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL
  Day 1 | 289.2 (14)
  Day 4 | 337.6 (15)

10. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) on Day 1 & 4 of Avibactam
Description: as for outcome 9
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL
  Day 1 | 47.29 (15)
  Day 4 | 49.59 (18)

11. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the End of the Dosing Interval (τ), Where τ=6 Hours (AUCtau) on Day 4 of Aztreonam
Description: AUCtau was defined as area under the concentration-time profile from time 0 to time tau. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL | 285.2 (14)

12. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the End of the Dosing Interval (τ), Where τ=6 Hours (AUCtau) on Day 4 of Avibactam
Description: as for outcome 11
Time Frame: Post dose on day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL | 44.41 (16)

13. Primary Outcome: Total Daily Area Under the Plasma Concentration-Time Profile From Time 0 to 24 Hours at Steady-State (AUC24,ss) on Day 4 of Aztreonam
Description: AUC24,ss was defined as total daily area under the plasma concentration-time profile from time 0 to 24 hours at steady-state. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL | 1142 (14)

14. Primary Outcome: Total Daily Area Under the Plasma Concentration-Time Profile From Time 0 to 24 Hours at Steady-State (AUC24,ss) on Day 4 of Avibactam
Description: as for outcome 13
Time Frame: Post dose on day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ug*hr/mL | 177.7 (16)

15. Primary Outcome: Renal Clearance (CLr) on Day 1 & 4 of Aztreonam
Description: CLr was calculated as cumulative amount of drug recovered unchanged in urine during the dosing interval (Ae) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau). AUCtau was defined as area under the concentration-time profile from time 0 to time tau. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre per hour (L/hr)
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
litre per hour (L/hr)
  Day 1: number analyzed (Participants) | 11
  Day 1 | 4.277 (14)
  Day 4 | 4.487 (23)

16. Primary Outcome: Renal Clearance (CLr) on Day 1 & 4 of Avibactam
Description: as for outcome 15
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre per hour (L/hr)
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
litre per hour (L/hr)
  Day 1: number analyzed (Participants) | 11
  Day 1 | 12.09 (18)
  Day 4 | 12.65 (25)

17. Secondary Outcome: Terminal Elimination Half-Life (T1/2) on Day 1 & 4 of Aztreonam
Description: Plasma terminal elimination half-life (T1/2) is the time measured for the plasma concentration to decrease by one half at the terminal phase.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
hours
  Day 1 | 1.890 (0.16597)
  Day 4 | 1.886 (0.20304)

18. Secondary Outcome: Terminal Elimination Half-Life (T1/2) on Day 1 & 4 of Avibactam
Description: as for outcome 17
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
hours
  Day 1 | 2.003 (0.34613)
  Day 4 | 4.061 (0.59180)

19. Secondary Outcome: Apparent Volume of Distribution at Steady-State (Vss) on Day 1 & 4 of Aztreonam
Description: Apparent volume of distribution (Vz) was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss was the Vz at steady-state. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Liter
  Day 1 | 13.69 (15)
  Day 4 | 12.81 (15)

20. Secondary Outcome: Apparent Volume of Distribution at Steady-State (Vss) on Day 1 & 4 of Avibactam
Description: Vz was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss was the Vz at steady-state. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Liter
  Day 1 | 21.36 (14)
  Day 4 | 17.96 (16)

21. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz) on Day 1 & 4 of Aztreonam
Description: Vz was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Liter
  Day 1 | 14.09 (16)
  Day 4 | 14.22 (16)

22. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz) on Day 1 & 4 of Avibactam
Description: as for outcome 21
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Liter
  Day 1 | 30.14 (22)
  Day 4 | 65.41 (26)

23. Secondary Outcome: Clearance (CL) on Day 1 & 4 of Aztreonam
Description: CL was a quantitative measure of the rate at which a drug substance was removed from the body. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre per hour (L/hr)
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
litre per hour (L/hr)
  Day 1 | 5.188 (14)
  Day 4 | 5.261 (14)

24. Secondary Outcome: Clearance (CL) on Day 1 & 4 of Avibactam
Description: as for outcome 23
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre per hour (L/hr)
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
litre per hour (L/hr)
  Day 1 | 10.56 (15)
  Day 4 | 11.26 (16)

25. Secondary Outcome: Time of Observed Maximum Plasma Concentration (Tmax) on Day 1 & 4 of Aztreonam
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
hours
  Day 1 | 2.92 [2.00 to 2.95]
  Day 4 | 2.92 [2.92 to 2.92]

26. Secondary Outcome: Time of Observed Maximum Plasma Concentration (Tmax) on Day 1 & 4 of Avibactam
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: Post dose on day 1 and day 4
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
hours
  Day 1 | 2.44 [2.00 to 2.95]
  Day 4 | 2.46 [2.00 to 2.92]

27. Secondary Outcome: Accumulation Ratio for Cmax (Rac,Cmax) on Day 4 of Aztreonam
Description: Accumulation ratio based on maximum plasma concentration (Rac,cmax) was calculated as: Rac,Cmax = Cmax at steady state (Day 4) divided by Cmax at first dose (Day 1). The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ratio | 1.149 (5)

28. Secondary Outcome: Accumulation Ratio for Cmax (Rac,Cmax) on Day 4 of Avibactam
Description: as for outcome 27
Time Frame: Post dose on day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ratio | 1.006 (7)

29. Secondary Outcome: Accumulation Ratio for AUCτ Following Multiple Dosing (Rac) on Day 4 of Aztreonam
Description: Rac was obtained from AUCtau at steady state (Day 4) divided by AUCtau after single dose (Day 1). AUCtau was defined as area under the concentration-time profile from time 0 to time tau. The geometric coefficient of variation is expressed in percentage.
Time Frame: Post dose on day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ratio | 1.204 (6)

30. Secondary Outcome: Accumulation Ratio for AUCτ Following Multiple Dosing (Rac) on Day 4 of Avibactam
Description: as for outcome 29
Time Frame: Post dose on day 4
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
ratio | 1.049 (6)

31. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse event (TEAE) means event between first dose of study treatment and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of death; inpatient hospitalization; life-threatening experience; disability; congenital anomaly or deemed significant for any other reason. Symptoms of infusion-related reactions (IRRs) may include, but were not limited to, fever, chills, flushing, hypotension, dyspnea, wheezing, back pain, abdominal pain, and urticaria. Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: From the first dose of study treatment to the last dose of study treatment date +28 +7 days (up to 2 months)
Population: The safety analysis set included all healthy Chinese participants who received at least one dose of investigational product (ATM-AVI).
Measure: Count of Participants; unit: Participants
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Participants
  Participants with treatment-emergent adverse events (all-causality) | 2
  Participants with treatment-emergent adverse events (treatment-related) | 1

32. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Criteria for vital signs abnormalities: increase or decrease from baseline in supine Systolic Blood Pressure (SBP) >=30 mm Hg and increase or decrease from baseline in supine Diastolic Blood Pressure (DBP) >=20 mm Hg.
Time Frame: From the first dose of study treatment to the last dose of study treatment date +28 +7 days (up to 2 months)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Participants
  Supine Diastolic Blood Pressure (mmHg): Change >= 20 mmHg increase from baseline | 0
  Supine Systolic Blood Pressure (mmHg): Change >= 30 mmHg increase from baseline | 0
  Supine Diastolic Blood Pressure (mmHg): Change >= 20 mmHg decrease from baseline | 0
  Supine Systolic Blood Pressure (mmHg): Change >= 30 mmHg decrease from baseline | 0

33. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs)
Description: ECG categorical summarization criteria: 1. PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): a) greater than or equal to (>=) 300 millisecond (msec), b) >=25% increase when baseline is > 200 msec or >=50% increase when baseline is less than or equal to (<=) 200 msec.
  2. QRS duration (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): a) >=140 msec, b) >=50% increase from baseline.
  3. QTcF interval (QT corrected using the Fridericia formula): a) >450 msec and <=480 msec, b) >480 msec and <=500 msec, c) >500 msec, d) >30 msec and <=60 msec increase from baseline, e) >60 msec increase from baseline.
Time Frame: From the first dose of study treatment to the last dose of study treatment date +28 +7 days (up to 2 months)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Participants
  PR INTERVAL NOT OTHERWISE SPECIFIED (msec): %Change >= 25/50% | 0
  QRS INTERVAL NOT OTHERWISE SPECIFIED (msec): %Change >= 50% | 0
  QTCF - FRIDERICIA'S CORRECTION FORMULA NOT OTHERWISE SPECIFIED (msec): 30 < Change <= 60 | 0
  QTCF - FRIDERICIA'S CORRECTION FORMULA NOT OTHERWISE SPECIFIED (msec): Change > 60 | 0

34. Secondary Outcome: Number of Participants With Abnormal Laboratory Assessments
Description: Following laboratory parameters were assessed against pre-defined abnormality criteria: hematology (basophils); clinical chemistry (urate); urinalysis (urine hemoglobin, nitrite, urine erythrocytes).
Time Frame: From the first dose of study treatment to the last dose of study treatment date +28 +7 days (up to 2 months)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
Number analyzed (Participants) | 12
Participants
  HEMATOLOGY: Basophils (10^3/mm^3) > 1.2x upper limit of normal (ULN) | 1
  CLINICAL CHEMISTRY: Urate (mg/dL) > 1.2x ULN | 1
  URINALYSIS: URINE Hemoglobin >= 1 | 3
  URINALYSIS: URINE Erythrocytes >= 20: number analyzed (Participants) | 4
  URINALYSIS: URINE Erythrocytes >= 20 | 2

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment to the last dose of study treatment date +28 +7 days (up to 2 months)
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | AZTREONAM-AVIBACTAM (ATM-AVI)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZTREONAM-AVIBACTAM (ATM-AVI) (N=12)
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04973826/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT04973826/SAP_001.pdf